CLINICAL TRIAL: NCT00882362
Title: Long-Term Administration Study of Aripiprazole as an Adjunctive Therapy in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 031-08-002; JapinCTI-090725
Record Dates: First submitted 2009-04-02; First posted 2009-04-16 (Estimated); Results first posted 2014-02-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2013-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: OPC-14597 (Aripiprazole)

INTERVENTIONS:
Drug: OPC-14597 (Aripiprazole) — administered orally once daily, 3 to 15 mg daily, 52 weeks

SUMMARY:
To examine the safety and efficacy of long term administration of aripiprazole as an adjunctive therapy, co-administered with either a selective serotonin reuptake inhibitor (SSRI) or a selective-norepinephrine reuptake inhibitor (SNRI), in subjects with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are either inpatients or outpatients
2. Patients who have the ability to understand and to provide informed consent to the examination, observation, and evaluation processes specified in this protocol, and have signed the informed consent form based on a full understanding of the trial
3. Patients diagnosed as having either "296.2x Major Depressive Disorder, Single Episode" or "296.3x Major Depressive Disorder, Recurrent" according to DSM-IV-TR, and for whom the current episode of major depressive disorder has been ongoing for more than 8 weeks.

Exclusion Criteria:

1. Female patients of child bearing potential who wish to become pregnant during the treatment period, or within 4 weeks after study completion/discontinuation
2. Female patients who are pregnant, possibly pregnant, or breast feeding
3. Patients judged to be unable to tolerate any type of antidepressant treatment (including drugs not being used in the current episode of major depressive disorder), based on treatment history to date
4. Patients who have previously received electro-convulsive therapy
5. Patients who have participated in clinical studies on medical devices or other drugs within the past month
6. Patients at risk of having serious adverse events or developing symptoms that could interfere with safety and efficacy evaluations (such as symptoms of fibromyalgia syndrome overlapping with symptoms of depression), based on previous medical history
7. Patients with a history or a complication of diabetes
8. Patients with thyroid disease (excluding patients who are stabilized on drug therapy for at least 3 months)
9. Patients with a history of serotonin syndrome or psychotropic neuroleptic malignant syndrome
10. Patients with a history of seizure disorder (epilepsy etc.)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2009-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — OPC-J
Locations (8):
- Japan (8):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuing Subjects: Subjects receiving the study drug for at least 4 weeks during the placebo-controlled double-blind treatment period of the 031-08-001 study
- Newly Entering Subjects: Newly entering elderly patients with major depressive disorder, aged 65 and above
Period: Overall Study
Arm/Group | Continuing Subjects | Newly Entering Subjects
Started | 122 | 33
Completed | 73 | 10
Not Completed | 49 | 23
Not completed — Adverse Event | 13 | 10
Not completed — Withdrawal by Subject | 13 | 10
Not completed — Lack of Efficacy | 3 | 0
Not completed — Protocol Violation | 7 | 2
Not completed — Pregnancy | 1 | 0
Not completed — Physician Decision | 5 | 1
Not completed — Diabetic glucose level or HbA1C>=6.5% | 2 | 0
Not completed — change of residence or other commitments | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuing Subjects | Newly Entering Subjects | Total
Number analyzed (Participants) | 122 | 33 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (8.6) | 73.1 (5.6) | 46.3 (16.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 122 | 0 | 122
  >=65 years | 0 | 33 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 23 | 78
  Male | 67 | 10 | 77
Region of Enrollment [Number; unit: participants]
  Japan | 122 | 33 | 155

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Change from baseline to Last Observation Carried Forward (LOCF).
  Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
  The questionnaire includes questions on the following symptoms
  1. Apparent sadness 2. Reported sadness 3. Inner tension 4. Reduced sleep 5. Reduced appetite 6. Concentration difficulties 7. Lassitude 8. Inability to feel 9. Pessimistic thoughts 10. Suicidal thoughts
Time Frame: Baseline(Day 1), Week52 or at discontinuation
Measure: Mean (Standard Error); unit: Rating Score
Arm/Group | Continuing Subjects | Newly Entering Subjects
Number analyzed (Participants) | 122 | 33
Rating Score | -4.60 (0.8) | -10.5 (1.9)

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Continuing Subjects | Newly Entering Subjects
Serious Adverse Events (participants affected / at risk) | 2/122 | 4/33
Other Adverse Events (participants affected / at risk) | 111/122 | 29/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuing Subjects (N=122) | Newly Entering Subjects (N=33)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haematoma Subdural (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1)
Abortion Missed (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuing Subjects (N=122) | Newly Entering Subjects (N=33)
Constipation (Gastrointestinal disorders) | 7 (9) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 9 (13) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Salivary Hypersecretion (Gastrointestinal disorders) | 2 (2) | 2 (3)
Nausea (Gastrointestinal disorders) | 7 (8) | 1 (1)
Oedema (General disorders) | 1 (1) | 2 (2)
Malaise (General disorders) | 6 (6) | 2 (3)
Nasopharyngitis (Infections and infestations) | 42 (62) | 5 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 3 (4) | 4 (7)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 4 (6)
Akathisia (Nervous system disorders) | 34 (39) | 8 (10)
Somnolence (Nervous system disorders) | 14 (15) | 5 (5)
Tremor (Nervous system disorders) | 12 (14) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 3 (3)
Dizziness Postural (Nervous system disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 6 (6) | 2 (3)
Dyskinesia (Nervous system disorders) | 7 (7) | 2 (2)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 6 (6) | 4 (4)
Major Depression (Psychiatric disorders) | 9 (10) | 1 (1)
Weight Increased (Investigations) | 39 (39) | 2 (2)
Blood Triglycerides Increased (Investigations) | 11 (13) | 1 (2)
Alanine Aminotransferase Increased (Investigations) | 9 (9) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 2 (2) | 2 (2)
Blood Creatine Phosphokinase Increased (Investigations) | 3 (3) | 2 (2)
Weight Decreased (Investigations) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No